CLINICAL TRIAL: NCT01693406
Title: Breast Milk and Infant Growth and Body Composition Among Healthy Mothers, Obese Mothers, and Mothers With Diabetes
Brief Title: Breast Milk and Infant Growth Among Lean, Overweight and Diabetic Mothers
Acronym: MIG
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Thrasher Research Fund (Other); American Diabetes Association (Other)
Responsible Party: Sponsor
Other Study IDs: 12-0629
Record Dates: First submitted 2012-09-21; First posted 2012-09-26 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Obesity; Type 2 Diabetes; Gestational Diabetes
Keywords: human milk; infant growth; obesity; diabetes; breastfeeding
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Diabetes, Gestational; Diabetes Mellitus; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human Milk, Plasma, Urine and Stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Normal Weight: Normal weight and normoglycemic women: Pre-pregnancy BMI between 18.5 - 24.9 kg/m2.
- Overweight/Obese: Overweight and normoglycemic women: Pre-pregnancy BMI between > 25 kg/m2.
- Gestational Diabetes: Women who develop gestational diabetes and return to normal glucose control after delivery.
- Type 2 Diabetes: Women who are overweight and have Type 2 Diabetes that was diagnosed before pregnancy: Pre-pregnancy BMI > 25 kg/m2.

SUMMARY:
Childhood obesity is a critical global public health concern. Breastfeeding is the ideal choice for infant nutrition. However, rapid and excess weight gain during infancy predicts later, even among breastfed infants. This risk is higher if mothers are obese and/or diabetic. Composition of bioactive components of breast milk may differ based between mothers who are normal weight (NW), overweight, or who have diabetes. Obesity and Type 2 Diabetes are associated with overall increases in inflammation and oxidative stress, but how breast milk composition is affected remains unknown. The investigators overarching goal is to determine how maternal obesity and Type 2 Diabetes impacts human breast milk composition and how differences in composition may impact infant growth and fat development. The investigators are undertaking a study that follows 20 Normal Weight, 20 Obese, 20 Gestational Diabetic, and 20 Type 2 Diabetic mothers and their infants over the first 4 months of life. The investigators will track infant weight and fat gain and monitor maternal glucose control. The investigators will also collect breast milk samples over the first 4 months and measure concentrations of growth and appetite hormones, cytokines, markers of oxidative stress and nutrient composition in milk. The investigators predict that concentrations of growth-regulatory hormones (insulin and leptin) in addition to the inflammatory cytokines and markers of oxidative stress will be lowest in breast milk from NW mothers, higher in breast milk from obese and gestational diabetic mothers, and highest in Type 2 Diabetic mothers' breast milk. The investigators expect these differences will be most pronounced in the first 2 weeks after birth. The investigators also predict that breast milk concentrations of these biomarkers will be associated with infant fat gain. What the investigators find will help understand how early infant nutrition and growth may affect that child's later risk of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Between 28-40 weeks gestation
* Plan to Exclusively Breastfeed for at least 5 months
* Between 20 - 35 years old
* Carrying a singleton pregnancy
* Parity less than or equal to 5
* Pre-pregnancy BMI between 18.5 and 39.9

Exclusion Criteria:

* No known infant anomalies or birth defects
* Maternal Type 1 Diabetes
* Maternal major medical condition (ie: Kidney Disease or Pre-eclampsia)
* Delivery of the infant before 35 weeks gestation
* Smoking During pregnancy

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will recruit pregnant women in the Denver Colorado area who plan to deliver their infant at the University of Colorado Hospital, and plan to exclusively breastfeed their infant for at least 5 months.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2012-08; Primary Completion 2020-08 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Change in infant percent body fat from birth to 4 months | Birth, 2 weeks, 1, 2, 3, and 4 months
  Body composition is measured by skin folds and air displacement plethysmography (PeaPod)

SECONDARY OUTCOMES:
Change in Human Milk Hormone Composition | 2 weeks, 1, 2, 3, and 4 months
  The investigators will analyze: insulin, leptin, adiponectin, and ghrelin concentrations in human milk samples collected at these time points
Change in Human Milk cytokine content | 2 weeks, 1, 2, 3, and 4 months
  The investigators will analyze: IL-10, IL-6, IL-8, and TNF-alpha concentrations in human milk samples collected at these time points
Change in Antioxidant capacity of human milk | 2 weeks, 1, 2, 3, and 4 months
  The investigators will analyze: TBARS, 8-OH-dG, HNE, and F2-isoprostane concentrations and total antioxidant capacity in human milk samples collected at these time points.

OTHER OUTCOMES:
Change in Human Milk Nutrient Composition | 2 weeks, 1, 2, 3, and 4 months
  The investigators will analyze: glucose, percent fat, protein and caloric content of human milk samples collected at these time points.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy F Krebs, MD, MS, Principal Investigator — University of Colorado, Denver; Linda A Barbour, MD, MSPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Derived] Odiase E, Frank DN, Young BE, Robertson CE, Kofonow JM, Davis KN, Berman LM, Krebs NF, Tang M. The Gut Microbiota Differ in Exclusively Breastfed and Formula-Fed United States Infants and are Associated with Growth Status. J Nutr. 2023 Sep;153(9):2612-2621. doi: 10.1016/j.tjnut.2023.07.009. Epub 2023 Jul 26. PMID 37506974
- [Derived] Lemas DJ, Young BE, Baker PR 2nd, Tomczik AC, Soderborg TK, Hernandez TL, de la Houssaye BA, Robertson CE, Rudolph MC, Ir D, Patinkin ZW, Krebs NF, Santorico SA, Weir T, Barbour LA, Frank DN, Friedman JE. Alterations in human milk leptin and insulin are associated with early changes in the infant intestinal microbiome. Am J Clin Nutr. 2016 May;103(5):1291-300. doi: 10.3945/ajcn.115.126375. PMID 27140533